CLINICAL TRIAL: NCT03748264
Title: User Preference/Validation Evaluation of the New Philips Respironics Positive Airway Pressure Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Respironics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ST-1203-APP-MS
Record Dates: First submitted 2018-11-13; First posted 2018-11-20 (Actual); Results first posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Sleep Disordered Breathing
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Standard of Care (Active Comparator): In the standard of care or the control condition, participants will receive the sites therapy initiation standard of care for setting up and educating the participants on their Obstructive Sleep Apnea, mask, and device information. This group will use a wireless modem that is attached to the PAP device and uploads adherence and other therapy information daily to a secured database (Encore Anywhere). With this method, therapy information is not directly available to the participant. Therapy information is available continuously to site staff personnel in the standard care arm.
  Interventions: Other: Standard of Care
- DreamMapper Application (Experimental): The DreamMapper Application group will receive the site's therapy initiation standard of care for setting up and educating the participants on their Obstructive Sleep Apnea, mask, and device information. Participants in this group will also download the DreamMapper application on their iPhone or Android smart phone. Therapy information and educational material will be available continuously to the participant with DreamMapper through the application. Study personnel will have access to adherence and therapy information continuously as well
  Interventions: Device: DreamMapper Application
- DreamMapper Application with Therapist Assist (Experimental): The DreamMapper Application wit Therapist Assist group will not receive the site's therapy initiation standard of care but will review the Therapist Assist automated educational material on Obstructive Sleep Apnea, and their Philips Respironics mask. and DreamMapper. These participants will download the DreamMapper application onto their iPhone or Android smart phone. Therapy information and educational material will be available continuously to the participant with DreamMapper. Study personnel will have access to adherence and therapy information continuously as well
  Interventions: Device: DreamMapper Application with Therapist Assist

INTERVENTIONS:
Other: Standard of Care — In the standard of care or the control condition, participants will receive the sites therapy initiation standard of care for setting up and educating the participants on their Obstructive Sleep Apnea, mask, and device information. This group will use a wireless modem that is attached to the PAP device and uploads adherence and other therapy information daily to a secured database (Encore Anywhere). With this method, therapy information is not directly available to the participant but will continuously be available to site staff personnel.
  Arms: Standard of Care
Device: DreamMapper Application — The DreamMapper application condition will receive the site's therapy initiation standard of care and will also download the DreamMapper application on their iPhone or Android smart phone. Therapy information and educational material will be available continuously to the participant with DreamMapper through the application. Study personnel will have access to adherence and therapy information continuously.
  Arms: DreamMapper Application
Device: DreamMapper Application with Therapist Assist — The DreamMapper with Therapist Assist will review the Therapist Assist automated educational material on Obstructive Sleep Apnea, their Philips Respironics mask and DreamMapper. These participants will download the DreamMapper application onto their iPhone or Android smart phone. Therapy information and educational material will be available continuously to the participant with DreamMapper. Study personnel will have access to adherence and therapy information continuously.
  Arms: DreamMapper Application with Therapist Assist

SUMMARY:
This pilot study is intended to evaluate the acceptance and performance of the DreamMapper application and the Therapist Assist educational tool in naïve patients with Obstructive Sleep Apnea who have been prescribed Positive Airway Pressure therapy. A total of approximately 60 naïve participants will be recruited.

DETAILED DESCRIPTION:
This is a randomized prospective trial designed to obtain subjective and objective feedback in a home use environment with participants using a Philips Respironics System One Positive Airway Pressure device. Participants will be randomly assigned to one of three methods of therapy introduction and monitoring:

1. Group 1: The first group, the control condition, participants will receive the sites therapy initiation standard of care for setting up and educating the participants on their Obstructive Sleep Apnea, mask, and device information. This group will use a wireless modem that is attached to the Positive Airway Pressure device and uploads adherence and other therapy information daily to a secured database (Encore Anywhere). With this method, therapy information is not directly available to the participant. Therapy information is available continuously to site staff personnel in the standard care arm.
2. Group 2: The second group will receive the site's therapy initiation standard of care for setting up and educating the participants on their Obstructive Sleep Apnea, mask, and device information. Participants in this group will also download the DreamMapper application on their iPhone or Android smart phone. Therapy information and educational material will be available continuously to the participant with DreamMapper through the application. Study personnel will have access to adherence and therapy information continuously as well.
3. Group 3: The third group will not receive the site's therapy initiation standard of care but will review the Therapist Assist automated educational material on Obstructive Sleep Apnea, and their Philips Respironics mask. and DreamMapper. These participants will download the DreamMapper application onto their iPhone or Android smart phone. Therapy information and educational material will be available continuously to the participant with DreamMapper. Study personnel will have access to adherence and therapy information continuously as well.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-75
* Diagnosis of Obstructive Sleep Apnea (OSA) with an Apnea Hypopnea Index (AHI) of at least 15 events/hour of sleep and a Central Apnea Index (CAI) ≤ 5 events /hour or ≤ 50% of the AHI.
* Newly diagnosed and Continuous Positive Airway Pressure (CPAP) Naïve.
* Currently owns and uses apps on an Android or iPhone smart phone.
* Willing to undergo an attended in lab Polysomnography (PSG)
* Willing and able to provide informed consent.
* Speaks and reads English as their primary language.

Exclusion Criteria:

* Presence of poorly managed or unstable major medical or psychiatric conditions that would interfere with the demands of the study, adherence to positive airway pressure, or the ability to complete the study. For example, unstable congestive heart failure, chronic lung disease with daytime hypercapnia, neuromuscular disease, psychiatric disease, cancer, or chronic renal failure.
* Participants who are unwilling to try Positive Airway Pressure (PAP) therapy.
* Participants currently prescribed oxygen therapy (as needed, nocturnal, or continuous).
* Participants with previously diagnosed respiratory failure or respiratory insufficiency.
* Recent surgery of the upper airway, noise, sinus, or eyes.
* Participant is prescribed a BiPAP device
* Commercial Drivers
* Shift workers
* Participants with untreated periodic limb movement syndrome, or restless legs syndrome (PLM Arousal Index > 15).
* Participants with untreated known diagnosis of Insomnia (score of 15-21(moderate severity) per Insomnia Severity Index (ISI) )
* Known diagnosis of bipolar disorder
* Participant with unstable anti- depressant medication (not stable for 3 months)

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-10-21 (Actual); Primary Completion 2014-05-27 (Actual); Study Completion 2014-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Wylie, MD, Principal Investigator — Arkansas Center For Sleep Medicine; Shalini Manchandra, MD, Principal Investigator — Program Director, Sleep Medicine Fellowship; Sukhdev Grover, MD, Principal Investigator — Sleep Center of Greater Pittsburgh; Eric Powell, PhD, Principal Investigator — Sleep Therapy & Research Center; Alan Lankford, MD, Principal Investigator — Sleep Disorders Center of Georgia, Inc.
Locations (5):
- United States (5):
  - Paul Wylie, MD, Little Rock, Arkansas
  - Sleep Disorders Center of Georgia, Inc., Atlanta, Georgia
  - Shalini Manchanda, MD, Indianapolis, Indiana
  - Sleep Center of Greater Pittsburgh, Pittsburgh, Pennsylvania
  - Sleep Therapy & Research Center, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care: All participants enrolled in to the Standard of care.
- DreamMapper Application: All participants that were enrolled into the DreamMapper Application.
- DreamMapper Application With Therapist Assist: All participants that were enrolled into the DreamMapper Application With Therapist Assist.
Period: Overall Study
Arm/Group | Standard of Care | DreamMapper Application | DreamMapper Application With Therapist Assist
Started | 21 | 21 | 20
Completed | 21 | 21 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard of Care: All participants that were enrolled into the Standard of Care.
- Total: Total of all reporting groups
Arm/Group | Standard of Care | DreamMapper Application | DreamMapper Application With Therapist Assist | Total
Number analyzed (Participants) | 21 | 21 | 20 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (11.4) | 46.9 (11.1) | 47.3 (10.0) | 47.0 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 11 | 28
  Male | 13 | 12 | 9 | 34
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 21 | 20 | 62
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 37.8 (8.5) | 36.4 (6.6) | 33.7 (5.1) | 36.0 (7.0)

OUTCOME MEASURES:

1. Primary Outcome: User Preference of the New Philips Respironics Positive Airway Pressure Application as Measured by the Attitudes Toward Use Questionnaire
Description: Participants will complete the Attitudes Toward Use Questionnaire (0 to 10 scale) to determine user preference of the New Philips Respironics Positive Airway Pressure Application. The higher the value the higher participant confidence.
Time Frame: 90 days
Population: All participants completed the study but not all participants completed the questionnaire for day 90. 6 standard of care participants did not complete the survey, 3 dreammapper and 1 dreammapper application with therapy assist did not complete the survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care | DreamMapper Application | DreamMapper Application With Therapist Assist
Number analyzed (Participants) | 15 | 18 | 19
units on a scale | 7.5 (3.6) | 7.9 (2.6) | 8.8 (1.5)

2. Secondary Outcome: Adherence
Description: Adherence will be measured among the three groups to determine which participants used their Positive Airway Pressure device most throughout the trial: DreamMapper compared to site standard of care compared to using DreamMapper and Therapist Assist.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: days per week
Arm/Group | Standard of Care | DreamMapper Application | DreamMapper Application With Therapist Assist
Number analyzed (Participants) | 21 | 21 | 20
days per week | 4.6 (2.4) | 4.8 (1.7) | 4.0 (2.5)

3. Secondary Outcome: Treatment Outcomes - Epworth Sleepiness Scale
Description: Treatment outcomes will be assess by the Epworth Sleepiness Scale. The Epworth Sleepiness is 8 question survey asking questions about likelihood to fall asleep, each questions is answered on a 0 to 3 scale, 0-no chance, 3-high chance, the higher the score the higher likelihood of daytime sleepiness. The scale is 0-24, 0-no chance to fall asleep.
Time Frame: 90 days
Population: All participants completed the study but not all participants completed the questionnaire for day 90. 5 standard of care participants did not complete the survey, 2 dreammapper and 1 dreammapper application with therapy assist did not complete the survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care | DreamMapper Application | DreamMapper Application With Therapist Assist
Number analyzed (Participants) | 16 | 19 | 19
units on a scale | 6.4 (4.0) | 7.9 (6.1) | 7.7 (4.8)

4. Secondary Outcome: Treatment Outcomes - Functional Outcomes of Sleep Questionnaire (FOSQ)
Description: Treatment outcomes will be assess by the Functional Outcomes of Sleep Questionnaire. The FOSQ is a specific quality of life questionnaire to determine functional status in adults; measures are designed to assess the impact of disorders of excessive sleepiness on multiple activities of everyday living and the extent to which these abilities are improved by effective treatment. It asks sets of questions for activity level, vigilance, intimacy and sexual relationships, general productivity, social outcome, rate the difficulty of performing a given activity on a 4-point scale (4-no difficulty to 1-extreme difficulty 0-I do not do it for other reasons). 10 questions are asked with the lowest score of 0 and the highest of score of 40. The lower the score the more difficulty it is to complete tasks.
Time Frame: 90 days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care | DreamMapper Application | DreamMapper Application With Therapist Assist
Number analyzed (Participants) | 16 | 19 | 19
units on a scale | 15.9 (4.4) | 16.0 (4.0) | 17.6 (2.0)

5. Secondary Outcome: Site Economic Savings Assessed by Number of Phone Calls.
Description: Site economics savings will be collected and analyzed by reviewing the number of phone calls per arm. Exact numeric amounts of savings are not available but number of calls is.
Time Frame: 90 days
Measure: Number; unit: number of phone calls
Arm/Group | Standard of Care | DreamMapper Application | DreamMapper Application With Therapist Assist
Number analyzed (Participants) | 21 | 21 | 20
number of phone calls | 6 | 7 | 9

6. Secondary Outcome: Patient Interactions
Description: Site and patient interactions will be assessed after 90 days by reviewing the exact number of unscheduled visits in each arm.
Time Frame: 90 days
Measure: Number; unit: number of unscheduled visits
Arm/Group | Standard of Care | DreamMapper Application | DreamMapper Application With Therapist Assist
Number analyzed (Participants) | 21 | 21 | 20
number of unscheduled visits | 2 | 3 | 4

7. Secondary Outcome: Mask Refits
Description: Number of patient visits requiring mask refits will be measured and recorded. The exact number of mask refits will be provided.
Time Frame: 90 days
Measure: Number; unit: number of refits
Arm/Group | Standard of Care | DreamMapper Application | DreamMapper Application With Therapist Assist
Number analyzed (Participants) | 21 | 21 | 20
number of refits | 2 | 2 | 3

8. Secondary Outcome: Overall Economic Cost Saving
Description: Analysis will be done on the overall economic cost savings from Therapist Assist and DreamMapper
Time Frame: 90 days
Population: Unable to be analyzed based upon site confidential information.
Arm/Group | Standard of Care | DreamMapper Application | DreamMapper Application With Therapist Assist
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 90 days
Groups:
- Standard of Care: In the standard of care or the control condition, participants will receive the sites therapy initiation standard of care for setting up and educating the participants on their Obstructive Sleep Apnea, mask, and device information. This group will use a wireless modem that is attached to the PAP device and uploads adherence and other therapy information daily to a secured database (Encore Anywhere). With this method, therapy information is not directly available to the participant. Therapy information is available continuously to site staff personnel in the standard care arm.Standard of Care: In the standard of care or the control condition, participants will receive the sites therapy initiation standard of care for setting up and educating the participants on their Obstructive Sleep Apnea, mask, and device information. This group will use a wireless modem that is attached to the PAP device and uploads adherence and other therapy information daily to a secured database (Encore Anywhere). With this method, therapy information is not directly available to the participant but will continuously be available to site staff personnel.
- DreamMapper: The DreamMapper Application group will receive the site's therapy initiation standard of care for setting up and educating the participants on their Obstructive Sleep Apnea, mask, and device information. Participants in this group will also download the DreamMapper application on their iPhone or Android smart phone. Therapy information and educational material will be available continuously to the participant with DreamMapper through the application. Study personnel will have access to adherence and therapy information continuously as wellDreamMapper Application: The DreamMapper application condition will receive the site's therapy initiation standard of care and will also download the DreamMapper application on their iPhone or Android smart phone. Therapy information and educational material will be available continuously to the participant with DreamMapper through the application. Study personnel will have access to adherence and therapy information continuously.
- DreamMapper Application With Therapist Assist: The DreamMapper Application wit Therapist Assist group will not receive the site's therapy initiation standard of care but will review the Therapist Assist automated educational material on Obstructive Sleep Apnea, and their Philips Respironics mask. and DreamMapper. These participants will download the DreamMapper application onto their iPhone or Android smart phone. Therapy information and educational material will be available continuously to the participant with DreamMapper. Study personnel will have access to adherence and therapy information continuously as wellDreamMapper Application with Therapist Assist: The DreamMapper with Therapist Assist will review the Therapist Assist automated educational material on Obstructive Sleep Apnea, their Philips Respironics mask and DreamMapper. These participants will download the DreamMapper application onto their iPhone or Android smart phone. Therapy information and educational material will be available continuously to the participant with DreamMapper. Study personnel will have access to adherence and therapy information continuously.
Arm/Group | Standard of Care | DreamMapper | DreamMapper Application With Therapist Assist
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/21 | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 7/21 | 4/21 | 4/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=21) | DreamMapper (N=21) | DreamMapper Application With Therapist Assist (N=20)
Influenza (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=21) | DreamMapper (N=21) | DreamMapper Application With Therapist Assist (N=20)
Irritated nostrils (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Weight Gain (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dry Upper Airway (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2)
Nasal irritation (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Adult Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Common Cold (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Right Ear Infection (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Broken bone right 4th finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Impression on face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pressure Sore (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No